CLINICAL TRIAL: NCT06078579
Title: Salivary and Serum Leptin Levels in Oral Lichen Planus Patients: A Case-Control Study.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bahaa Mahmoud Fawzy El Nomrosy, Dentist, Cairo University
Other Study IDs: 20723
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Oral Lichen Planus; Leptin Levels
Keywords: salivary; Serum
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — ELISA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral lichen planus patients: Assessment of salivary and serum leptin levels
  Interventions: Diagnostic Test: Leptin
- Healthy control group: Assessment of salivary and serum leptin levels
  Interventions: Diagnostic Test: Leptin

INTERVENTIONS:
Diagnostic Test: Leptin — Assessment of salivary and serum leptin levels in oral lichen planus patients and healthy controls

SUMMARY:
This study aims to evaluate the levels of leptin in both saliva and serum samples of patients diagnosed with oral lichen.

DETAILED DESCRIPTION:
Oral lichen planus is a frequently encountered chronic muco-cutaneous condition with a high prevalence rate. The condition can be classified as an autoimmune disorder.Although the exact cause of this condition is unknown, some potential risk factors should be taken into account, such as systemic disorders, psychogenic diseases, dental restorations, and certain medications.

The oral lesions exhibit a mostly bilateral pattern, often manifesting in the inner buccal mucosa. The condition can be classified into three distinct forms, namely the reticular form, atrophic form, and bullous-erosive form.

The condition is classified as a premalignant lesion due to its significant likelihood of undergoing malignant transformation. The disease is characterized by the presence of T-lymphocyte infiltration in the basal cell layer of the epithelium and the presence of cytoid bodies, which are distinct histopathologic markers.

Leptin, a hormone generated by adipocytes, is involved in immunological responses and contributes to the development of autoimmunity. The presence of dyslipidemia has been found to be associated with lipoprotein (LP) abnormalities. Consequently, this study was undertaken to assess the blood leptin levels and lipid profile in individuals with LP. Leptin, a polypeptide hormone, is produced and released by white adipose tissue.

Multiple research have substantiated an increase in leptin levels among persons exhibiting elevated body mass index (BMI) and a higher percentage of total body fat. Additionally, it is involved in the cellular immune response and facilitates the development of autoimmunity.

There is a proposition suggesting that leptin has a role in the promotion of cytokine generation and modulation of helper T cells, potentially implicating its involvement in the pathogenesis of psoriasis. The available information about leptin status in dermatological illnesses other than psoriasis is currently sparse. It is plausible that it may have a significant role in the pathogenesis of lichen planus.

However, there is a lack of literature regarding the levels of leptin in LP. There is an association between dyslipidemia and LP. Numerous investigations have consistently demonstrated notable deviations in lipid profile levels between individuals with LP and those in normal, healthy control cohorts. These findings have led researchers to posit a correlation between chronic inflammation and dyslipidemia, hence heightening the susceptibility to cardiovascular illnesses.

The potential impact of leptin on the progression of LP is being investigated. The objective of this study was to conduct a comparative analysis of blood leptin levels between individuals recently diagnosed with LP and a control group consisting of healthy individuals. Additionally, an assessment was conducted to examine the correlation between leptin levels, lipid profile, and the length of illness.

ELIGIBILITY:
Inclusion Criteria:

* Ages for both sexes fall between 30 and 70.
* Symptomatic OLP has been diagnosed clinically and verified histologically.
* Participants who sign a written consent form after being fully informed about the study.

Exclusion Criteria:

* Treatment with a systemic or locally administered systemic medication within the previous three months before the commencement of the research.
* Patients now taking or who have just stopped taking an NSAIDs (both steroidal and non steroidal) for pain or inflammation.
* Patients who have been diagnosed with a malignant tumor or tumors.
* Women who are expecting or nursing.
* Inmates, the mentally ill, the elderly, etc, all fall into this category.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OLP patients and healthy controls were selected will be selected from "out-patient clinic" of Oral Medicine, Periodontology and Oral Diagnosis Department ;Faculty of Dentistry, Cairo university and from "out-patient" of Boulak El Dakroor general hospital.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weam Ah Rashwan, PHD, Study Director — Cairo University; Olfat Ga Shaker, PHD, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Aryanian Z, Shirzadian A, Hatami P, Dadras H. High Incidence of Metabolic Syndrome Components in Lichen Planus Patients: A Prospective Cross-Sectional Study. Int J Clin Pract. 2022 Jan 31;2022:7184678. doi: 10.1155/2022/7184678. eCollection 2022. PMID 35685585
- [Background] Matarese G, Moschos S, Mantzoros CS. Leptin in immunology. J Immunol. 2005 Mar 15;174(6):3137-42. doi: 10.4049/jimmunol.174.6.3137. PMID 15749839
- Available data/document: Study Protocol — https://www.ijhsr.org/IJHSR_Vol.5_Issue.10_Oct2015/20.pdf — www.researchgate.net/publication/344178013_Serum_Leptin_and_Lipid_Profile_in_Lichen_Planus_A_case_control_study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process has taken 1 year, starting from December 2023 till December 2024; all recruitment processes were done in the Cairo University outpatient clinic.
Pre-assignment Details: There is no washout that has been done; some of the enrolled participants were excluded because they were currently on systemic steroid medication or taking topical steroids for lesions.
Groups:
- Oral Lichen Planus Patients: Assessment of salivary and serum leptin levels
  Leptin: Assessment of salivary and serum leptin levels in oral lichen planus patients
- Healthy Control Group: Assessment of salivary and serum leptin levels
  Leptin: Assessment of salivary and serum leptin healthy controls
Period: Overall Study
Arm/Group | Oral Lichen Planus Patients | Healthy Control Group
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Lichen Planus Patients | Healthy Control Group | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 38 | 69
  >=65 years | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.77 (13.37) | 34.51 (12.53) | 42.641 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 13 | 18 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 39 | 39 | 78
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 28.47 (3.95) | 28.77 (3.32) | 28.62 (3.62)

OUTCOME MEASURES:

1. Primary Outcome: Serum Leptin Level
Description: Assessment of serum leptin levels in in oral lichen planus patients
Time Frame: Baseline
Population: Levels of leptin in serum of patients with active oral lichen planus
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Serum Leptin Levels in OLP Patients: Leptin levels in serum of patients with active oral lichen planus disease
- Serum Leptin Levels in Healthy Control Subjects: Serum leptin levels measurement in healthy control subjects
Arm/Group | Serum Leptin Levels in OLP Patients | Serum Leptin Levels in Healthy Control Subjects
Number analyzed (Participants) | 39 | 39
ng/ml | 13.23 (7.29) | 4.20 (1.23)

2. Secondary Outcome: Salivary Leptin Levels
Description: Assessment of salivary leptin levels in oral lichen planus patients
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Salivary Leptin Levels in OLP Patients: Salivary leptin levels measurement in patients with active oral lichen planus disease
- Salivary Leptin Levels in Healthy Control Subjects: Salivary leptin levels measurment in healthy control subjects
Arm/Group | Salivary Leptin Levels in OLP Patients | Salivary Leptin Levels in Healthy Control Subjects
Number analyzed (Participants) | 39 | 39
ng/ml | 15.31 (6.59) | 4.90 (1.26)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 3 months following the intervention
Description: There are no serious risk events because the trial is simple: taking saliva or taking a blood sample is easy, and none of this can cause mortality.
Groups:
- Oral Lichen Planus Patients: Patients with active symptomatic oral lichen planus
- Healthy Control Subjects: Healthy controls that not have any active aystemic disease
Arm/Group | Oral Lichen Planus Patients | Healthy Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT06078579/Prot_SAP_002.pdf